CLINICAL TRIAL: NCT01090063
Title: An Investigator-Initiated, Open-label Study Evaluating the Efficacy and Safety of Ustekinumab in Patients With Moderate to Severe Palmar Plantar Psoriasis
Brief Title: Efficacy and Safety of Ustekinumab in Patients With Moderate to Severe Palmar Plantar Psoriasis
Acronym: PPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Palmar Plantar Psoriasis
Record Dates: First submitted 2010-03-15; First posted 2010-03-19 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Moderate to Severe Palmar Plantar Psoriasis
Keywords: Palmar Plantar Psoriasis
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ustekinumab — Dosing will consist of a 45mg subcutaneous injection for patients weighing less than 100 kg and a 90 mg subcutaneous injection for patients whose weight is greater than 100 kg. Dosing will begin on week 0 followed by subsequent dosing on week 4 and week 16.
  Other Names: Stelara

SUMMARY:
The purpose of this study is to determine the short and long term safety and effectiveness of ustekinumab in subjects with moderate to severe chronic palmar plantar psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 18 and 85 years of age with palmar plantar psoriasis with well defined psoriatic plaques on the palms and/or soles with a Physician Global Assessment (PGA) of 3 or higher who are unresponsive to topical management. Pustules, fissures and psoriatic arthritis may be present but are not required.
2. Adults in general good health as determined by the Investigator based upon the results of medical history, laboratory profile, and physical examination.
3. Females of reproductive potential are eligible to participate in the study if they have a negative urine pregnancy test at screening and baseline and who are using 2 forms of effective birth control.
4. Palmar/Plantar PGA of 3 or more

Exclusion Criteria:

1. Psoriasis patients without palm and/or sole psoriasis or a palmar/plantar PGA score of less than 3
2. Patients younger than 18 and older than 85 years old.
3. Evidence of skin conditions at the time of the screening visit (e.g. eczema) other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis
4. Receipt of any investigational drugs within 4 weeks of study drug initiation
5. Psoralens + UltraViolet A (PUVA) or oral systemic treatments within 4 weeks of study drug initiation.
6. Biologics within 3 months of study initiation
7. Ultraviolet B (UVB) therapy or topical steroids within 2 weeks of study drug initiation
8. A prior history of tuberculosis, and/or a positive Purified Protein Derivative (PPD) skin test/Chest X-Ray (CXR) at screening without appropriate treatment. Treatment of latent Tuberculosis (TB) infections (for those with positive PPD tests) must be initiated prior to therapy.
9. Receipt of live vaccines 1 month prior to or while in study
10. Chronic hepatitis B or hepatitis C infection
11. History of alcohol or drug abuse one year before and during the study.
12. Known Human Immunodeficiency Virus (HIV)-positive status or any other immune-suppressing disease.
13. Any grade 3 or 4 adverse event, or laboratory toxicity, at the time of the screening visit or at any time during the study
14. Presence of a grade 3 or 4 infection <30 days prior to the screening visit, between the screening visit and the first day of treatment on study, or any time during the study that in the opinion of the Investigator would preclude participation in the study.
15. Any internal malignancy within 5 years (fully excised cutaneous, basal cell carcinoma or squamous cell carcinoma are exceptions)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice B Gottlieb, MD, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from Apr 2010 to Sept 2011 in the dermatology clinic of a tertiary care hospital.
Pre-assignment Details: Washout of 2 weeks for topicals, 4 weeks for all other biologics and systemics prior to baseline dosage.
Groups:
- Main: All participants were treated the same
Period: Screen
Arm/Group | Main
Started | 28
Completed | 24
Not Completed | 4
Not completed — Screen Failed | 4
Period: Treatment
Arm/Group | Main
Started | 24
Completed | 20
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Main
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving a Palmar/Plantar PGA Score of 0 or 1 at Week 16.
Time Frame: 16 weeks
Population: Number of participants completing enrollment. Lost values carried forward as last observation carried forward
Measure: Number; unit: percentage of participants
Groups:
- Main: Percentage of patients achieving a palmar/plantar PGA score of 0 or 1 at week 16.
Arm/Group | Main
Number analyzed (Participants) | 24
percentage of participants | 0.375

2. Secondary Outcome: PGA Score Over Time From Baseline to Week 24
Description: Measurement of subject's palmar and plantar psoriasis severity as measured by the Physician's Global Assessment (PGA) scale, which rates the severity of psoriasis using the measures of erythema, scaling and induration. Scores are from 0 to 4, in 1 unit increments. A score of 4 is very severe, and a score of 0 is clear.
Time Frame: Baseline, 24 weeks
Population: All participants who enrolled. Early terminations were carried as last observation carried forward.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Median PGA: Median PGA at Week 24
Arm/Group | Median PGA
Number analyzed (Participants) | 24
units on a scale | 2.5 (1.4) [0 to 4]

3. Secondary Outcome: Pustule Count (if Present at Baseline) From Baseline to Week 24
Description: Number of pustules present in each subject
Time Frame: Baseline, 24 weeks
Population: All participants who enrolled. Early terminations were carried as last observation carried forward.
Measure: Mean (Standard Deviation); unit: pustules
Groups:
- Mean Pustule Count at Baseline: Average number of pustules present in all subjects at baseline
- Mean Pustule Count at Week 24: Average number of pustules present in all subjects at week 24
Arm/Group | Mean Pustule Count at Baseline | Mean Pustule Count at Week 24
Number analyzed (Participants) | 24 | 24
pustules | 8.2 (19.7) | 13.2 (28.0)

4. Secondary Outcome: Fissure Count (if Present at Baseline) From Baseline to Week 24
Description: Number of discrete fissures on the hands and feet of each subject.
Time Frame: Baseline, 24 weeks
Population: All participants who enrolled. Early terminations were carried as last observation carried forward.
Measure: Mean (Standard Deviation); unit: fissures
Groups:
- Mean Baseline Fissure Count: Average number of fissures found on hands and feet at baseline
- Mean Week 24 Fissure Count: Average number of fissures found on hands and feet at Week 24
Arm/Group | Mean Baseline Fissure Count | Mean Week 24 Fissure Count
Number analyzed (Participants) | 24 | 24
fissures | 3.5 (5.5) | 3.7 (6.8)

5. Secondary Outcome: Pruritus Visual Analog Scale From Baseline to Week 24
Description: Patient's score on the questionnaire of "how itchy are you", as measured in mm from the left end of scale. Maximum score is 100, minimum score is 0. 100 indicates maximum itch (worse outcome), 0 indicates minimum itch (better outcome).
Time Frame: Baseline, 24 weeks
Population: All participants who enrolled. Early terminations were carried as last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Baseline Pruritus VAS Score: Average pruritus VAS score as measured at baseline. Maximum score is 100, minimum score is 0. 100 indicates maximum itch (worse outcome), 0 indicates minimum itch (better outcome).
- Mean Week 24 Pruritus VAS Score: Average pruritus VAS score as measured at week 24. Maximum score is 100, minimum score is 0. 100 indicates maximum itch (worse outcome), 0 indicates minimum itch (better outcome).
Arm/Group | Mean Baseline Pruritus VAS Score | Mean Week 24 Pruritus VAS Score
Number analyzed (Participants) | 24 | 24
units on a scale | 47.9 (33.4) | 30 (31.9)

6. Secondary Outcome: Pain Visual Analog Scale From Baseline to Week 24
Description: Patient's score on the questionnaire of "how much pain are you experiencing from your disease of your hands and feet", as measured in mm from the left end of scale. Maximum score is 100, minimum score is 0. Visual Analog Scale (VAS). 100 indicates maximum pain (worse outcome), 0 indicates minimum pain (better outcome).
Time Frame: Baseline, 24 weeks
Population: All participants who enrolled. Early terminations were carried as last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Baseline Pain VAS Score: Average score of the pain VAS at baseline. 100 indicates maximum pain (worse outcome), 0 indicates minimum pain (better outcome).
- Mean Week 24 Pain VAS Score: Average score of the pain VAS at Week 24. 100 indicates maximum pain (worse outcome), 0 indicates minimum pain (better outcome).
Arm/Group | Mean Baseline Pain VAS Score | Mean Week 24 Pain VAS Score
Number analyzed (Participants) | 24 | 24
units on a scale | 50.9 (34.3) | 30.8 (30.9)

7. Secondary Outcome: Safety Outcome Measures
Description: All adverse events (AE's) will be recorded and monitored. At each of the study visits, patients will be questioned about the occurrence of new AE's since the last visit, or the outcome of any AE's that were reported at previous visits. Upon study completion of the first 10 subjects the principal investigator will review all adverse events to check for trends.
Time Frame: 24 weeks
Population: All participants who enrolled. Participants terminating prior to week 24 had their data carried forward as lost to follow-up.
Measure: Number; unit: participants
Arm/Group | Number of Participants With AEs
Number analyzed (Participants) | 24
participants | 17

ADVERSE EVENTS:
Arm/Group | Main
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 6/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main (N=24)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Mild Self-Limited Upper Respiratory Infection
Acneiform Eruption (Skin and subcutaneous tissue disorders) | 2 (2) — Mild Acneiform Eruption, Self Limited

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No